CLINICAL TRIAL: NCT00763243
Title: Pilot Study of the Feasibility and Efficacy of Working Memory Training in Children With Cochlear Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0808-01B
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Results first posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-04

CONDITIONS: Bilateral Hearing Loss
Keywords: profound bilateral hearing loss with cochlear implants
MeSH Terms: conditions — Hearing Loss, Bilateral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cogmed Working Memory Training (Experimental): Cogmed Working Memory Training Program
  Interventions: Behavioral: Cogmed Working Memory Training Program

INTERVENTIONS:
Behavioral: Cogmed Working Memory Training Program — The Cogmed Working Memory Training program is a 5-week program of computer-based exercises that require the user to complete tasks involving verbal, visual, or combined verbal-visual memory skills. In addition to memory skills, Cogmed tasks demand attention, concentration, and reasoning skills. Users are expected to practice Cogmed exercises at home for 40 minutes/day, 5 days/week, during the 5-week training period. The program uses an adaptive algorithm that presents users with problems of increasing difficulty at a level slightly higher than that at which they have recently achieved success.
  Other Names: Cogmed

SUMMARY:
This study is an investigation of the effect of a computer-based working memory training program on memory and language processing in at-risk children (e.g., those with working memory weaknesses) who have received cochlear implants.

DETAILED DESCRIPTION:
The long-term goal of this research program is to improve speech-language outcomes in prelingually deaf children who receive CIs. The objective of this proposal is to investigate the short-term effects of a novel working memory training program on memory, learning, and speech-language outcomes in children with CIs. The specific hypothesis of this project is that completion of a behaviorally-based training program designed to increase working memory capacity will improve attention, working memory span, and working memory-related speech-language processing in a group of deaf children with CIs. This hypothesis is based on past research demonstrating the efficacy of working memory training programs in improving attention and working memory in children with attention deficits, as well as on past research showing an association between working memory and speech-language outcomes in children with CIs. Knowledge about the effects of working memory training on CI speech-language outcomes will provide a better understanding of the process by which children with CIs learn speech-language following implantation and may offer an entirely new avenue of intervention to improve speech-language outcomes, particularly in deaf children who show limited improvement following implantation.

The specific aims of this study are:

1. Specific Aim 1: Determine the feasibility and application of a novel, computer-based working memory training program when applied to children with CIs. We hypothesize that children with CIs will show a progression of learning in both auditory and visual working memory during the training program that will mirror that of normal-hearing children.
2. Specific Aim 2: Determine the effect of the working memory training program on core attention, concentration, and working memory processes of children with CIs. We hypothesize that children with CIs will show improvement on both laboratory-based and parent-report measures of attention, concentration, and working memory processes after working memory training, compared to a baseline period.
3. Specific Aim 3: Determine the effect of the working memory training program on working memory-related speech-language outcome measures in children with CIs. We hypothesize that children with CIs will show improvement on auditory working memory, verbal naming fluency, and word repetition after training.

ELIGIBILITY:
Inclusion Criteria:

* age 7-16 years at the time of study enrollment,
* profound bilateral hearing loss (> 90 dB HL in the better hearing ear),
* implantation prior to age 3 years,
* use of multichannel CI's,
* a monolingual English home environment,
* enrollment in an aural rehabilitative program that encourages the development of speaking and listening skills,
* educational environment that uses oral or total communication (TC) strategies,
* sufficient speech perception and language competence to complete basic word and sentence repetition tasks,
* no significant developmental delay or neurological condition that, in the opinion of the investigators, would interfere markedly with cognitive functioning,
* Windows-based PC at home capable of running Cogmed working memory training software,
* mild or greater deficit in working memory, as shown by either (a) a Behavior Rating Inventory of Executive Function (BRIEF) working memory T-score of 50 or higher or (b) a Digit Span scaled score of 10 or lower. Subjects will be discontinued if during the study they have any new or changed intervention (including medication) that involves working memory, attention, concentration, or executive functioning.

Exclusion Criteria:

* Under 7 years or over 16 years of age at time of study entry
* Implantation after age 3 years
* Bilingual or non-English-speaking home environment
* Primary use of American Sign Language (ASL)

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2008-08; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William G. Kronenberger, PhD, Principal Investigator — Indiana University
Locations (1):
- Riley Hospital for Children, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited over a 2 year period from a database of families whose children had received cochlear implants at a large university-based teaching hospital and who had consented to be contacted for participation in research studies.
Pre-assignment Details: All eligible subjects were assigned to Cogmed working memory training.
Groups:
- Cogmed Working Memory Training: Cogmed Working Memory Training Program
  Cogmed Working Memory Training Program : The Cogmed Working Memory Training program is a 5-week program of computer-based exercises that require the user to complete tasks involving verbal, visual, or combined verbal-visual memory skills. In addition to memory skills, Cogmed tasks demand attention, concentration, and reasoning skills. Users are expected to practice Cogmed exercises at home for 40 minutes/day, 5 days/week, during the 5-week training period. The program uses an adaptive algorithm that presents users with problems of increasing difficulty at a level slightly higher than that at which they have recently achieved success.
Period: Waiting Period
Arm/Group | Cogmed Working Memory Training
Started | 9
Completed | 9
Not Completed | 0
Period: Training Period
Arm/Group | Cogmed Working Memory Training
Started | 9
Completed | 9
Not Completed | 0
Period: 1-Month Follow-Up Period
Arm/Group | Cogmed Working Memory Training
Started | 9
Completed | 9
Not Completed | 0
Period: 6-Month Follow-Up Period
Arm/Group | Cogmed Working Memory Training
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cogmed Working Memory Training
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.2 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Digit Span Total Raw Score (Construct Measured: Verbal Short-Term/Working Memory)
Description: This is a measure of digit span forward and digit span backward based on the WISC-III Digit span subtest. Subjects are presented with sequences of single digits, starting with 2 digits, which increase by 1 digit after 2 sequences are presented at each digit length. The test is discontinued when 2 items are missed at the same digit length. Raw score is the number of items (digit sequences) answered correctly. Subjects must recall all digits either in forward (digit span forward) or backward (digit span backward) order. The Digit Span test is a measure of verbal short-term/working memory. Scores range from 0 to 28, with higher scores indicating better verbal short-term/working memory.
Time Frame: Administered at Screening Visit, Pretraining Visit (2-5 weeks later), Posttraining Visit (5 weeks after Pretraining Visit), 1 month follow-up visit (1 month after Posttraining Visit), and 6 month follow-up visit (6 months after Posttraining Visit)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Screening Visit: Screening Visit at Study Entry
  Cogmed Working Memory Training Program : The Cogmed Working Memory Training program is a 5-week program of computer-based exercises that require the user to complete tasks involving verbal, visual, or combined verbal-visual memory skills. In addition to memory skills, Cogmed tasks demand attention, concentration, and reasoning skills. Users are expected to practice Cogmed exercises at home for 40 minutes/day, 5 days/week, during the 5-week training period. The program uses an adaptive algorithm that presents users with problems of increasing difficulty at a level slightly higher than that at which they have recently achieved success.
- Pretraining Visit: Visit that occurs 2-5 Weeks after Screening Visit (at the end of the Waiting Period) and immediately before Cogmed WMT started
- Posttraining Visit: Visit that occurs immediately after 5-week Cogmed working memory training (end of Training Period)
- 1-Month Follow Up Visit: Visit 1 month after Cogmed working memory training was completed
- 6-Month Follow Up Visit: Visit 6 months after Cogmed working memory training completed
Arm/Group | Screening Visit | Pretraining Visit | Posttraining Visit | 1-Month Follow Up Visit | 6-Month Follow Up Visit
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9
Scores on a scale | 11 (3.28) | 11.22 (2.54) | 12.89 (2.93) | 13 (3.64) | 11.56 (2.79)
Statistical Analysis 1: Comparison: Screening Visit vs Pretraining Visit; Change during waiting period (no intervention); no change was hypothesized; Test type: Superiority or Other; p = 0.766, t-test, 2 sided; t(8)=0.31; Mean Difference (Final Values) = 0.22, 95% CI 2-sided [-1.44 to 1.89], Standard Deviation 2.17
Statistical Analysis 2: Comparison: Pretraining Visit vs Posttraining Visit; Change during the training period; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; t(8)=5.0; Mean Difference (Final Values) = 1.67, 95% CI 2-sided [0.90 to 2.44], Standard Deviation 1.0
Statistical Analysis 3: Comparison: Pretraining Visit vs 1-Month Follow Up Visit; Change from pre-training through follow-up period; Test type: Superiority or Other; p = 0.021, t-test, 2 sided; t(8)=2.87; Mean Difference (Final Values) = 1.78, 95% CI 2-sided [0.35 to 3.20], Standard Deviation 1.86
Statistical Analysis 4: Comparison: Pretraining Visit vs 6-Month Follow Up Visit; Change from pretraining to 6 month follow up; Test type: Superiority or Other; p = 0.40, t-test, 2 sided; t(8)=0.89; Mean Difference (Final Values) = 0.33, 95% CI 2-sided [-0.53 to 1.19], Standard Deviation 1.12

2. Primary Outcome: Spatial Span Total Raw Score (Construct Measured: Visuospatial Short-Term/Working Memory)
Description: This is a measure of memory for sequential spatial locations (forward and backward), based on the subject touching one of 10 blocks in the same sequence (forward) or in the reverse sequence (backward) that they were touched by the examiner. This subtest is based on the WISC-IV-Integrated Spatial Span subtest. The examiner points to blocks on a board, sequentially, starting with a sequence of two blocks (locations), which increase by 1 block (location) after 2 sequences are presented at each span length. The test is discontinued when 2 items are missed at the same spatial span length. Raw score is the number of items (complete sequences) answered correctly. The Spatial Span test is a measure of visuospatial short-term/working memory. Scores range from 0 to 28, with higher scores indicating better visuospatial short-term/working memory.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Screening Visit | Pretraining Visit | Posttraining Visit | 1-Month Follow Up Visit | 6-Month Follow Up Visit
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9
Scores on a scale | 13 (2.24) | 14.33 (3.35) | 16.78 (3.83) | 16.44 (4.13) | 15.11 (4.26)
Statistical Analysis 1: Comparison: Screening Visit vs Pretraining Visit; Change during waiting period of no intervention; Test type: Superiority or Other; p = 0.11, t-test, 2 sided; t(8)=1.79; Mean Difference (Final Values) = 1.33, 95% CI 2-sided [-0.39 to 3.05], Standard Deviation 2.24
Statistical Analysis 2: Comparison: Pretraining Visit vs Posttraining Visit; Change during training period; Test type: Superiority or Other; p = 0.004, t-test, 2 sided; t(8)=4.05; Mean Difference (Final Values) = 2.44, 95% CI 2-sided [1.05 to 3.84], Standard Deviation 1.81
Statistical Analysis 3: Comparison: Pretraining Visit vs 1-Month Follow Up Visit; 1 Month Follow Up change from pre-training; Test type: Superiority or Other; p = 0.072, t-test, 2 sided; t(8)=2.07; Mean Difference (Final Values) = 2.11, 95% CI 2-sided [-0.24 to 4.46], Standard Deviation 3.06
Statistical Analysis 4: Comparison: Pretraining Visit vs 6-Month Follow Up Visit; 6 month follow up change from pre-training; Test type: Superiority or Other; p = 0.34, t-test, 2 sided; t(8)=1.02; Mean Difference (Final Values) = 0.78, 95% CI 2-sided [-0.97 to 2.53], Standard Deviation 2.28

3. Primary Outcome: Behavior Rating Inventory of Executive Function (BRIEF) - Working Memory Subscale Raw Score (Construct Measured: Behavioral Attention-Concentration and Working Memory)
Description: The BRIEF is a parent-report questionnaire of executive functioning behaviors in children. For each item, parents rate whether the child engages in the behavior "never" (=1), "sometimes" (=2), or "often" (=3). Raw scores for subscales are sums of item scores. The Working Memory subscale consists of 10 items asking about attention, concentration, and active controlled memory. Working Memory subscale raw scores are measures of attention, concentration, and working memory, and range from 10 to 30. Higher raw scores indicate more problems with attention, concentration, and working memory.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Screening Visit | Pretraining Visit | Posttraining Visit | 1-Month Follow Up Visit | 6-Month Follow Up Visit
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9
Scores on a scale | 16.89 (3.92) | 17.11 (3.72) | 15.33 (3.61) | 16.22 (3.93) | 16.44 (3.50)
Statistical Analysis 1: Comparison: Screening Visit vs Pretraining Visit; Waiting period - no treatment; Test type: Superiority or Other; p = 0.729, t-test, 2 sided; t(8)=0.36; Mean Difference (Final Values) = 0.22, 95% CI 2-sided [-1.20 to 1.65], Standard Deviation 1.86
Statistical Analysis 2: Comparison: Pretraining Visit vs Posttraining Visit; Training Period - Pretraining to Post-Training Visit; Test type: Superiority or Other; p = 0.039, t-test, 2 sided; t(8)=2.46; Mean Difference (Final Values) = -1.78, 95% CI 2-sided [-3.44 to -0.11], Standard Deviation 2.17
Statistical Analysis 3: Comparison: Pretraining Visit vs 1-Month Follow Up Visit; 1 Month Follow Up Period from Pretraining; Test type: Superiority or Other; p = 0.40, t-test, 2 sided; t(8)=0.90; Mean Difference (Final Values) = -0.89, 95% CI 2-sided [-3.17 to 1.40], Standard Deviation 2.98
Statistical Analysis 4: Comparison: Pretraining Visit vs 6-Month Follow Up Visit; 6 Month Follow Up period from pretraining; Test type: Superiority or Other; p = 0.40, t-test, 2 sided; t(8)=0.89; Mean Difference (Final Values) = -0.67, 95% CI 2-sided [-2.59 to 1.26], Standard Deviation 2.50

ADVERSE EVENTS:
Arm/Group | Screening Visit | Pretraining Visit | Posttraining Visit | 1-Month Follow Up Visit | 6-Month Follow Up Visit
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes